CLINICAL TRIAL: NCT00396331
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Safety and Efficacy of AMD3100 (240 µg/kg) Added to a G-CSF Mobilization Regimen in Poor Mobilizing Adult Patients Who Have Previously Failed Stem Cell Collection/Attempts
Brief Title: AMD3100 (Plerixafor) With G-CSF in Poor Mobilizing Adult Patients Who Previously Failed Hematopoietic Stem Cell (HSC) Collection/Attempts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD31002112
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Autologous Stem Cell Transplantation
Keywords: Multiple Myeloma; Non-Hodgkin's Lymphoma; autologous transplantation; AMD3100; stem cell mobilization; plerixafor
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-CSF plus Plerixafor (Experimental)
  Interventions: Drug: G-CSF plus plerixafor

INTERVENTIONS:
Drug: G-CSF plus plerixafor — Participants underwent mobilization with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days, administered by subcutaneous injection (SC) injection each morning. On the evening of Day 4, participants received a dose of plerixafor 240 µg/kg, administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF 10 µg/kg and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor (within 60 minutes after administration of G-CSF). Participants continued to receive an evening dose of plerixafor followed the next day by a morning dose of G-CSF and apheresis for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
  Other Names: AMD3100; Mozobil

SUMMARY:
This study evaluates the safety, efficacy, and pharmacokinetics (PK) of plerixafor given in addition to granulocyte-colony stimulating factor (G-CSF) for collection of peripheral blood stem cells (PBSCs) for autologous transplantation in patients who would benefit from an autologous stem cell transplant but have failed previous collections or collection attempts with a mobilization regimen of G-CSF alone, chemotherapy and G-CSF, or any other conventional therapy including cytokines, chemotherapy and cytokines and bone marrow harvests.

The only change to standard of care of a mobilization regimen that includes G-CSF is the addition of a dose of AMD3100 (plerixafor) on the evening prior to each day of apheresis.

Efficacy outcomes include quantification of CD34+ cells in the apheresis product and assessment of successful polymorphonuclear leukocyte (PMN) and platelet (PLT) engraftment after transplantation. PK outcomes include analysis of repeated doses of plerixafor.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, prospective, open-label study. Once 70 patients have enrolled, subsequent patients enrolled should have a diagnosis of lymphoma. Patients who would benefit from an autologous stem cell transplant, who have failed previous collections or collection attempts with a mobilization regimen of granulocyte colony-stimulating factor (G-CSF) alone, chemotherapy and G-CSF, or any other conventional therapy including cytokines, chemotherapy and cytokines and bone marrow harvests, and who meet the inclusion/exclusion criteria are eligible to receive plerixafor as outlined in this protocol. The only change to standard of care of a mobilization regimen that includes G-CSF is the addition of a dose of plerixafor on the evening prior to each day of apheresis.

Patients will undergo mobilization with G-CSF (10 µg/kg) for 4 days. On Day 4, plerixafor (240 µg/kg) will be administered in the evening prior to the first apheresis and each subsequent evening prior to apheresis thereafter, such that there is a 10 to 11 hour interval between dosing and the initiation of apheresis. Patients will continue to receive G-CSF on each day of apheresis. Patients will undergo a minimum of 2 and a maximum of 7 aphereses or until ≥2*10^6 CD34+ cells/kg are collected, whichever occurs first. In addition, the mobilization of NHL tumor cells and the pharmacokinetics of repeat doses of plerixafor will be examined.

After the last apheresis has been completed, or after the patient has collected ≥2*10^6 CD34+ cells/kg, he/she will be treated with high-dose chemotherapy in preparation for transplantation. Patients will be transplanted with cells obtained from the G-CSF with plerixafor mobilization regimen. In the event that the minimum number of ≥2*10^6 cells for transplantation are not obtained from the first mobilization with plerixafor, cells may be retained and pooled for transplantation with those from a second mobilization with plerixafor (or from prior mobilization with other agents), at the investigator's discretion. If a second mobilization with plerixafor is attempted, a minimum rest interval of one week should be allowed between the last apheresis of the first regimen and the first dose of G-CSF of the second. The number of CD34+ cells mobilized in the peripheral blood (PB), collected in the apheresis product, and the number of apheresis sessions performed will be measured. Success of the transplantation will be evaluated by the time to engraftment of polymorphonuclear leukocytes (PMN) and platelets (PLT). Participants will be assessed for durability of their transplant for 12 months after transplantation.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to undergo autologous transplantation
* Has failed previous collections or collection attempts with a mobilization regimen of granulocyte colony-stimulating factor (G-CSF), chemotherapy and G-CSF or any other conventional therapy including cytokines, chemotherapy and cytokines or bone marrow harvest.
* Eastern Co-operative Oncology Group (ECOG) performance status of 0 or 1
* ≥3 weeks since last cycle of chemotherapy (thalidomide, dexamethasone, and Velcade™ are not considered prior chemotherapy for the purpose of this study) NOTE: Although thalidomide, dexamethasone, and Velcade™ are not considered prior chemotherapy for the purpose of this study, none are to be administered within 7 days prior to the first dose of G-CSF (see Exclusion Criteria).
* The patient has recovered from all acute toxic effects of prior chemotherapy
* White blood cell count (WBC) >2.5*10^9/L
* Absolute neutrophil count >1.5*10^9/L
* Platelet count >85*10^9/L
* Serum creatinine ≤1.5 mg/dl
* Creatinine clearance >60 ml/min
* Aspartate aminotransferase (AST), alanine transaminase (ALT) and total bilirubin <2x upper limit of normal (ULN)
* Left ventricle ejection fraction >45% (by normal echocardiogram (ECHO) or multiple gated acquisition (MUGA) scan)
* Forced expiratory volume in one minute (FEV1) >60% of predicted or diffusion lung capacity for carbon monoxide (DLCO) ≥45% of predicted
* No active infection of hepatitis B or C
* Negative for HIV
* Signed informed consent
* Women of child-bearing potential agree to use an approved form of contraception

Exclusion Criteria:

* Once 70 patients have enrolled, patients with diagnoses other than lymphoma are not eligible (eg, acute myeloid leukemia, chronic lymphocytic leukemia, or multiple myeloma).
* A co-morbid condition which, in the view of the investigators, renders the patient at high risk from treatment complications
* A residual acute medical condition resulting from prior chemotherapy
* Received Neupogen™, thalidomide, dexamethasone, and/or Velcade™ within 7 days prior to the first dose of G-CSF
* Brain metastases or carcinomatous meningitis
* Acute infection
* Fever (temperature >38°C/100.4°F)
* Hypercalcaemia (>1 mg/dL above the ULN)
* Positive pregnancy test in female patients
* Lactating females
* Patients of child-bearing potential unwilling to implement adequate birth control
* Patients whose actual body weight exceeds 175% of their ideal body weight
* Patients who previously received experimental therapy within 4 weeks of enrolling in this protocol or who are currently enrolled in another experimental protocol during the Mobilization phase

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (8):
  - City of Hope National Medical Center', Duarte, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Blood & Marrow Transplant Group of Georgia, Atlanta, Georgia
  - University of Mississippi Medical Center, Div of Hematology, Jackson, Mississippi
  - Kansas City Cancer Centers, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin, Blood and Bone Marrow Transplant, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were enrolled in the study but never received plerixafor treatment so are not included below. Reasons for not receiving plerixafor included disease progression (2), infection (1) and insurance issues (1).
Groups:
- G-CSF Plus Plerixafor: Participants were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
Period: Overall Study
Arm/Group | G-CSF Plus Plerixafor
Started | 100
Number of Participants Treated | 100
Number of Participants Transplanted | 87 (7 participants had two transplants)
Completed | 68
Not Completed | 32
Not completed — Failed to mobilize - no transplant | 8
Not completed — Did not go on to transplant | 5
Not completed — Lost to Follow-up | 3
Not completed — Death | 16

BASELINE CHARACTERISTICS:
Groups:
- Non-Hodgkin's Lymphoma: Participants with non-Hodgkin's lymphoma (NHL) were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
- Hodgkin's Disease: Participants with Hodgkin's disease (HD) were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
- Multiple Myeloma: Participants with multiple myeloma (MM) were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
- Other Cancers: Participants with 'other' cancers (desmoplastic small round cell tumor, acute myeloid leukemia, and testicular cancer) were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
- Total: Total of all reporting groups
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | Total
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (10.0) | 45.6 (15.5) | 62.6 (11.3) | 32.7 (28.9) | 54.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 10 | 5 | 1 | 45
  Male | 37 | 11 | 5 | 2 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 60 | 17 | 9 | 3 | 89
  Black or African American | 3 | 1 | 1 | 0 | 5
  Asian | 2 | 1 | 0 | 0 | 3
  Hispanic/Latino | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Participant Counts Summarizing Adverse Events (AEs) During the Treatment Period
Description: Number of participants with adverse events (AEs) collected from Day 1 (start of G-CSF mobilization) to the day before starting chemotherapy. AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe, life-threatening) and relatedness to study treatment (5 point scale from 'not related' to 'definitely related').
Time Frame: Day 1 to approximately day 38
Population: Safety population of all participants who received at least 1 dose of plerixafor.
Measure: Number; unit: Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Participants
  Participants Reporting At Least 1 AE | 65 | 20 | 9 | 3 | 97
  Adverse Events by Severity -Mild | 42 | 12 | 7 | 1 | 62
  Adverse Events by Severity -Moderate | 18 | 8 | 1 | 0 | 27
  Adverse Events by Severity -Severe | 5 | 0 | 1 | 2 | 8
  Adverse Events by Severity -Life Threatening | 0 | 0 | 0 | 0 | 0
  AE Relationship to Study Drug -Not Related | 10 | 4 | 4 | 0 | 18
  AE Relationship to Study Drug-Probably Not Related | 8 | 2 | 1 | 0 | 11
  AE Relationship to Study Drug -Possibly Related | 16 | 4 | 1 | 0 | 21
  AE Relationship to Study Drug -Probably Related | 22 | 2 | 2 | 1 | 27
  AE Relationship to Study Drug -Definitely Related | 9 | 8 | 1 | 2 | 20

2. Primary Outcome: Proportion of Participants Who Achieved ≥2*10^6 CD34+ Cells/kg Following Treatment With Plerixafor and G-CSF
Description: Proportion of participants who reached the target of at least 2*10^6 CD34+ cells/kg collected during up to 7 aphereses.
Time Frame: Day 5 to Day 11 (up to 7 apheresis)
Population: Full analysis set of participants who received at least 1 dose of plerixafor. These results do not include results from the second course of plerixafor treatment and second course of apheresis for the 7 participants who had 2 courses of apheresis.
Measure: Number; unit: Proportion of Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Proportion of Participants | .773 | .714 | 1.00 | .667 | .780

3. Secondary Outcome: Median Number of Days to Polymorphonuclear Leukocyte (PMN) Engraftment
Description: The number of days from transplantation to successful engraftment as measured by PMN >=0.5*10^9 /L for 3 days or >=1.0*10^9 /L for 1 day.
Time Frame: approximately 2 months (1 month post transplant)
Population: Participants who received a transplant and had a successful PMN engraftment. Seven participants (4 with HD, 2 with MM, and 1 with testicular cancer) received a second transplant. Two transplants (1 in a participant with NHL and 1 in a participant with MM) did not result in PMN engraftment and are therefore not included in the analysis.
Measure: Median (Full Range); unit: Days
Units Other Than Participants: Transplants with PMN engraftment
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 60 | 16 | 8 | 1 | 85
Number analyzed (Transplants with PMN engraftment) | 60 | 20 | 10 | 2 | 92
Days | 12.0 [2.0 to 19.0] | 12.0 [11.0 to 15.0] | 13.0 [9.0 to 16.0] | 10.0 [7.0 to 13.0] | 12.0 [2.0 to 19.0]

4. Secondary Outcome: Median Number of Days to Platelet (PLT) Engraftment
Description: The number of days from transplantation to successful engraftment as measured by platelet value of >=20*10^9/L for 7 days without transfusion.
Time Frame: Approximately 2 months (1 month post transplant)
Population: Participants who received a transplant and had a successful PLT engraftment. Seven participants (4 with HD, 2 with MM, and 1 with testicular cancer) received a second transplant. Four transplants (2 in participants with NHL and 2 in participants with MM) did not result in PLT engraftment and are therefore not included in the analysis.
Measure: Median (Full Range); unit: Days
Units Other Than Participants: Transplants with PLT engraftment
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 59 | 16 | 7 | 1 | 83
Number analyzed (Transplants with PLT engraftment) | 59 | 20 | 9 | 2 | 90
Days | 21.0 [7.0 to 88.0] | 21.0 [15.0 to 81.0] | 19.0 [16.0 to 24.0] | 26.0 [3.0 to 49.0] | 21.0 [3.0 to 88.0]

5. Secondary Outcome: Number of Participants With Durable Engraftment 12 Months After Autologous Transplantation
Description: The number of participants maintaining a durable graft 12 months after transplantation. A durable graft was defined as maintenance of normal blood counts: PLT >50*10^9/L without transfusion for at least 2 weeks prior to the visit; hemoglobin level >= 10 g/dL with no erythropoietin or transfusions for at least 1 month prior to the visit; and absolute neutrophil count (ANC) > 1,000 (1*10^9/L) with no G-CSF for at least 1 week prior to the visit.
Time Frame: Approximately 13 months (12 months post transplant )
Population: Participants who received autologous stem cell transplantation and were evaluable 12 months post transplant. The 3 participants who did not have durable grafts included 2 participants whose PLT level never recovered to >50*10^9/L and 1 who had low hemoglobin at the 12-month visit.
Measure: Number; unit: Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 46 | 14 | 8 | 0 | 68
Participants | 44 | 14 | 7 |  | 65

6. Primary Outcome: Proportion of Participants Who Achieved ≥5*10^6 CD34+ Cells/kg Following Treatment With Plerixafor and G-CSF
Description: Proportion of participants who reached the target of at least 5*10^6 CD34+ cells/kg collected during up to 7 apheresis.
Time Frame: Day 5 to Day 11 (up to 7 aphereses)
Population: Full analysis set of participants who received at least 1 dose of plerixafor. These results do not include results from the second course of plerixafor treatment and second course of apheresis for the 7 participants who had two courses of apheresis.
Measure: Number; unit: Proportion of Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Proportion of Participants | 0.288 | 0.429 | 0.70 | 0.667 | 0.37

7. Secondary Outcome: Number of Participants With Non-Hodgkin's Lymphoma (NHL) Who Had Evidence of Tumor Cell Mobilization After G-CSF or Plerixafor Administration
Description: The number of participants with Bcl2 translocation in post-treatment samples.
Time Frame: Up to Day 7
Population: NHL participants with known follicular or transformed (follicular to diffuse large cell) lymphoma who provided samples for tumor cell mobilization analysis.
  Outcome is not reported because there were insufficient samples for analysis.
Arm/Group | Non-Hodgkin's Lymphoma
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Who Achieved ≥2*10^6 CD34+ Cells/kg Collected During Both Courses of Treatment With Plerixafor and G-CSF
Description: Number of participants who had at least 2*10^6 CD34+ cells/kg collected by apheresis during both the first and the second courses of treatment together.
Time Frame: Day 5 up to Month 6 (up to 7 aphereses in each course of treatment)
Population: Participants who received one course or two courses of plerixafor. Four NHL participants and 3 HD participants had two courses of plerixafor and the sum of CD34+ cells/kg collected in both courses is included.
Measure: Number; unit: Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Participants | 54 | 18 | 10 | 2 | 84

9. Secondary Outcome: Number of Participants Who Achieved ≥5*10^6 CD34+ Cells/kg Collected During Both Courses of Treatment With Plerixafor and G-CSF
Description: Number of participants who had at least 5*10^6 CD34+ cells/kg collected by apheresis during both the first and the second courses of treatment together.
Time Frame: Day 5 up to Month 6 (up to 7 aphereses in each course of treatment)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers | All Patients
Number analyzed (Participants) | 66 | 21 | 10 | 3 | 100
Participants | 21 | 9 | 7 | 2 | 39

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 4
Description: Maximum plasma concentration (Cmax) of plerixafor following daily doses of 240 µg/kg plerixafor, determined directly from the concentration-time data.
Time Frame: Day 4 (following first plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PK Subpopulation: Participants in the pharmacokinetic (PK) subpopulation that offered blood samples for PK analysis. Participants were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 7 aphereses or until ≥ 2*10^6 CD34+ cells/kg were collected.
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 19
ng/mL | 796 (305)

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) on Day 7
Description: as for outcome 10
Time Frame: Day 7 (following fourth plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 15
ng/mL | 894 (227)

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) on Day 4
Description: Time to maximum plasma concentration (Tmax) of plerixafor following daily doses of 240 µg/kg plerixafor, determined directly from the concentration-time data
Time Frame: Day 4 (following first plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 19
Hours | 0.500 [0.0500 to .750]

13. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) on Day 7
Description: as for outcome 12
Time Frame: Day 7 (following fourth plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 15
Hours | 0.500 [0.417 to 0.600]

14. Secondary Outcome: Area Under the Steady-state Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Sample (AUC0-last) on Day 4
Description: Area under the steady-state plasma concentration time curve from time zero to the last quantifiable sample after each plerixafor daily dose of 240 µg/kg, determined using the linear trapezoidal rule.
Time Frame: Days 4 -5 (following first plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 19
ng*h/mL | 4578 (1715)

15. Secondary Outcome: Area Under the Steady-state Plasma Concentration Time Curve From Time Zero to the Last Quantifiable Sample (AUC0-last) on Day 7
Description: as for outcome 14
Time Frame: Days 7-8 (following fourth plerixafor administration)
Population: Participants who provided blood samples for pharmacokinetic (PK) analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | PK Subpopulation
Number analyzed (Participants) | 15
ng*h/mL | 5496 (1339)

ADVERSE EVENTS:
Time Frame: First day of G-CSF mobilization to the day prior to chemotherapy/ablative treatment in preparation for the first transplant. This timeframe includes G-CSF and plerixafor administration, and the rest period.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Each AE table includes all events, regardless of reported relationship to study treatment or grade.
Arm/Group | Non-Hodgkin's Lymphoma | Hodgkin's Disease | Multiple Myeloma | Other Cancers
Serious Adverse Events (participants affected / at risk) | 4/66 | 0/21 | 1/10 | 1/3
Other Adverse Events (participants affected / at risk) | 64/66 | 20/21 | 9/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (N=66) | Hodgkin's Disease (N=21) | Multiple Myeloma (N=10) | Other Cancers (N=3)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Central line infection (Infections and infestations) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (N=66) | Hodgkin's Disease (N=21) | Multiple Myeloma (N=10) | Other Cancers (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 7 | 4 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 8 | 4 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 15 | 6 | 3 | 1
Paraesthesia oral (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0 | 1
Asthenia (General disorders) | 4 | 0 | 1 | 0
Catheter related complication (General disorders) | 1 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 1 | 0 | 0
Catheter site pain (General disorders) | 4 | 1 | 2 | 1
Catheter thrombosis (General disorders) | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 3 | 0 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 28 | 8 | 4 | 2
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Infusion site erythema (General disorders) | 2 | 0 | 0 | 0
Injection site discolouration (General disorders) | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 18 | 6 | 2 | 1
Injection site haematoma (General disorders) | 4 | 1 | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 1 | 0
Injection site inflammation (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 2 | 0 | 0 | 2
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 5 | 0 | 0 | 2
Injection site reaction (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 6 | 1 | 0 | 0
Pain (General disorders) | 7 | 3 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Blood culture positive (Investigations) | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0
Culture positive (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 2 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 3 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 17 | 7 | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Testicular choriocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 7 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 14 | 4 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 11 | 6 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 7 | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0
Dysphoria (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 3 | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 4 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Neovascularisation (Vascular disorders) | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees to submit the draft of any proposed public release or proposed publication to Genzyme and Genzyme may review the proposed public release or draft of the publication for up to 30 days prior to submission for public release, presentation or use. PI agrees (1) to withhold submission for an additional period not to exceed 60 days to allow Genzyme to take action to protect patent rights or trade secret rights (2) to give due consideration to any editorial comments of Genzyme.